CLINICAL TRIAL: NCT05856929
Title: Sexual Function and Reproductive Function of Kidney Transplant Recipients
Brief Title: Sexual Dysfunction After Renal Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20222236-C-1
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-09

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Renal transplant group
  Interventions: Other: no Intervention

INTERVENTIONS:
Other: no Intervention — no intervention

SUMMARY:
A questionnaire will be send to kidney transplant recipients to investigate characteristics of them and their sexual function, all participants in the survey are anonymous and voluntary, then analyse these characteristics.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone kidney transplantation for more than six months

Exclusion Criteria:

* having no sexual partner, being under 18 or over 70 years of age, exhibiting abnormal mental behavior, having poor understanding and communication ability, having low intelligence, or having a congenital sexual disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who have undergone kidney transplantation for more than six months
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the number of participants is up to 500 | 2024.06

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xijing Hospital, Xi'an, Shaanxi
  - Department of Urology, Xi'an

IPD SHARING:
Plan to Share IPD: No
no plan to share